CLINICAL TRIAL: NCT07004894
Title: Effects of Neuromuscular Reeducation Versus Friction Massage in Lateral Epicondylitis: A Randomized Control Trial
Brief Title: Effects of Neuromuscular Reeducation Versus Friction Massage in Lateral Epicondylitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Furqan Ahmed Siddiqi (Other)
Responsible Party: Sponsor-Investigator, Furqan Ahmed Siddiqi, Foundation University Islamabad, Foundation University Islamabad
Organization: Foundation University Islamabad (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/75
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-16 (Actual); Status verified 2024-07

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular reeducation (Experimental): Group A will recieve treatment of ultrasound followed by neuromuscular re-education+ strengthning exercises For the 1st two weeks; cross friction massage with active movement will be performed.
  For the next two weeks; longitudinal friction massage with active movement will be performed.
  Interventions: Procedure: Neuromuscular re-education(experimental)
- Friction massage (Active Comparator): Group B will receive standard treatment of ultrasound followed by friction massage+ strengthning exercises For the 1st two weeks; cross friction massage alone will be performed. For the last two weeks; longitudinal friction massage alone will be performed.
  Interventions: Procedure: Friction massage(standard protocol)

INTERVENTIONS:
Procedure: Neuromuscular re-education(experimental) — All participants will receive 4weeks of intervention with a frequency of 2-3 days/week with a period of rest in between. 5 minutes of ultrasound will be given followed by neuromuscular reeducation technique (5-10 minutes duration) which includes for the 1st two weeks; cross friction massage with active movement and for the last two weeks longitudinal friction massage with active movement will be performed and strengthening protocol will be given.
  The exercise protocol will be taught to the patient by an experienced physiotherapist and supervised on the subsequent sessions. The protocol will be gradually progressed as per the patient's tolerance.
  Arms: Neuromuscular reeducation
Procedure: Friction massage(standard protocol) — All participants will receive 4weeks of intervention with a frequency of 2-3 days/week with a period of rest in between. 5 minutes of ultrasound will be given followed by friction massage technique(5-10 minutes duration) which includes for the 1st two weeks; cross friction massage alone and for the last two weeks longitudinal friction massage alone will be performed and strengthening protocol will be given.
  The exercise protocol will be taught to the patient by an experienced physiotherapist and supervised on the subsequent sessions. The protocol will be gradually progressed as per the patient's tolerance.
  Arms: Friction massage

SUMMARY:
This study is a randomised control trial and the purpose of this study is to determine the effects of neuromuscular reeducation versus friction massage in lateral epicondylitis.

DETAILED DESCRIPTION:
Participants will be recruited into their respective groups using a coin toss method. Lateral epicondylitis will be assessed using the following tests:

Cozen's test Maudsley's test Mills test

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed cases of lateral epicondylitis
2. Age 25-50 years
3. Both genders
4. Postive tests; cozens, maudsley's, mills (at least any of 2)

Exclusion Criteria:

1. Recent elbow fractures or dislocations
2. Elbow joint instability
3. Active joint disease
4. Open wounds around elbow joints

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Lateral Epicondylitis Pain | Variable will be assessed at pre and post treatment for the total interval of 4 weeks.
  It will be measured using numeric pain rating scale (NPRS) in which the subjects select a number ranging from 0-10 according to their intensity of pain. '0' score indicates no pain while '10' indicates worst pain experienced.
Range of Motion | Variable will be assessed at pre and post treatment for the total interval of 4 weeks.
  Range of motion will be measured using goniometer. An instrument with movable and stationary arm used to measure range of motion at joint. It will be used to measure range of motion of flexion and extension at elbow joint, forearm pronation and supination, and flexion, extension, radial deviation, ulnar deviation at wrist joint.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan